CLINICAL TRIAL: NCT02833870
Title: Non-drug Taken Charge of Alzheimer's Disease: Profit Musical Activities
Brief Title: Non-pharmacological Care of Alzheimer's Disease: Benefice of Musical Interventions
Acronym: MusicAlzheimer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: PO13125 252Au12
Record Dates: First submitted 2016-07-08; First posted 2016-07-14 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Alzheimer's Disease (AD) and Related Disorders
MeSH Terms: conditions — Alzheimer Disease | interventions — Cooking; Methods

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (3):
- Musical intervention (Experimental)
  Interventions: Behavioral: Musical intervention
- Non-musical (cooking) intervention (Experimental)
  Interventions: Behavioral: Non-musical (cooking) intervention
- Control with no intervention (Active Comparator)
  Interventions: Behavioral: Control with no intervention

INTERVENTIONS:
Behavioral: Musical intervention
  Arms: Musical intervention
Behavioral: Non-musical (cooking) intervention
  Arms: Non-musical (cooking) intervention
Behavioral: Control with no intervention
  Arms: Control with no intervention

SUMMARY:
Cares of Alzheimer's disease (AD) and related disorders are presenting a real public health challenge. Because of the limited effectiveness of pharmacological treatments, there is a growing interest in care approach based on nonpharmacological treatments, such as musical interventions. Several lines of evidence suggest that musical interventions could improve behaviour, emotion and even cognition in patients with AD. However, very few studies respond to the methodological constraints required for clinical controlled trials carried out in well selected groups of patients. The efficiency of such care approaches is not scientifically proved yet and the impact of musical interventions has rarely been compared to another pleasant intervention, leaving open the question about the specific benefits of music in patients with dementia. The main goal of this research project is to demonstrate short and longer-term efficiencies and the specificity of musical interventions in dementia by investigating their effects not only in patients but also in familial and professional caregivers.

DETAILED DESCRIPTION:
To generalize previous results showing that non pharmacological therapy based on musical interventions improved emotional state in patients with severe AD to a larger sample of patients and to demonstrate the possible effects on caregivers, the investigators carried out a randomized controlled study with three parallel arms in institutionalized patients with severe AD (study 1) and in patients with mild AD leaving at home (study 2) to compare the impact of two interventions, a musical and a non-musical (cooking), to a control group (without any intervention). The control activity (cooking) was selected because it shares different features with music. Both interventions provide pleasure, are multisensory and may trigger old memories. In addition, both activities can be carried out in groups. A protocol consisting of various selected tests and questionnaires was used to assess the emotional, behavioural and cognitive abilities. Professional and familial caregivers also filled out other questionnaires to assess potential indirect benefits from both interventions on caregiver burnout and familial caregiver burden. Six assessments were proposed, two before, two during and two after interventions (follow-up) to respectively evaluate short and longer-term benefits of both interventions whereas test -retest effects will be controlled. Psychologists in charge to these assessments will be blind in regard to patients' group (musical versus cooking sessions, no intervention). Data were analyzed with methods from social psychology to decode non-verbal behaviours (e.g. visual contact) and emotional indexes in facial and verbal expressions and with methods from classical neuropsychology and from health domain. The collaboration between the two university teams from Lille and the special care unit (Pole EHPAD-USLD in Reims Hospital) provided complementary skills to this project that ensured its feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Older People and francophones living in institutions
* Presenting a cortical degenerative disease
* Male or female
* Age 60 to 99 years
* French Mother tongue
* People enjoying a social security scheme
* Patient Participation Agreement and of the person of trust or his legal representative.

Exclusion Criteria:

* Patients without cortical degenerative disease
* Patients with uncorrected profound hearing loss
* Not affiliated with a social security scheme Patients .
* Patients refusing to participate in the study or with the agreement of the person of trust or his legal representative was not obtained
* Patient protected by law

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Overall score in the Neuropsychiatric Inventory | up to 11 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France